CLINICAL TRIAL: NCT03092700
Title: Effects of Pulmonary Rehabilitation on Dyspnoea Affective Dimension and Emotional Cognition in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Pulmonary Rehabilitation, Dyspnoea and Emotional Cognition in COPD
Acronym: READ-COG BPCO
Status: Completed | Type: Observational
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00045-48
Record Dates: First submitted 2017-03-18; First posted 2017-03-28 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: COPD; Dyspnea; Rehabilitation; Tobacco Use; Emotional Disturbances
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Tobacco Use; Affective Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate whether pulmonary rehabilitation improves emotional cognition, using facial emotions recognition and smile production, by improving the emotional dimension of dyspnoea in patients with chronic obstructive pulmonary disease (COPD).To evaluate whether pulmonary rehabilitation improves emotional cognition, using facial emotions recognition and smile production, by improving the emotional dimension of dyspnoea in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The aim of the study will be to evaluate the effect of pulmonary rehabilitation on dyspnoea emotional component and on emotional cognition. It will add a better understanding of the mechanisms of pulmonary rehabilitation on dyspnoea.

Patients with COPD will be included before starting a pulmonary rehabilitation and be evaluated with questionnaires (including the Multidimensional Dyspnea Profile, and quality of life questionnaires), emotional cognition (at rest and right after an endurance test, using some short movies sequences and pictures of faces expressing some well defined emotions) and smile production analysis.

After having followed a pulmonary rehabilitation, the same evaluation will be realised and results will be compared before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with pulmonary rehabilitation indication, hospitalized in Department of Pulmonary Diseases in La Pitié-Salpêtrière, Paris, France.
* Age of 40 at least.

Exclusion Criteria:

* Facial paralysis
* Neuromuscular disease
* Contraindication for pulmonary rehabilitation
* Severe depression syndrom or psychiatric disease
* Drug use
* Impaired vision
* Higher functions disorders (Mini Mental Score Examination < 26)
* Severe obesity (BMI>40kg/m²)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted for a pulmonary rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
emotional cognition | 6 weeks
  Emotional cognition in patients with chronic dyspnoea using time to recognize some emotions on short movies and pictures of facial emotions.

SECONDARY OUTCOMES:
Correlation between physical improvement, quality of life improvement and time to recognize facial emotions. | 6 weeks
  Correlations
Correlations between physical improvement and production of the smile. | 6 weeks
  Correlations

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique Paris Est, Groupe Hospitalier Pitié-Salpêtrière, Paris, France